CLINICAL TRIAL: NCT00135798
Title: The Adult-to-adult Living Donor Liver Transplantation Cohort Study (A2ALL) Low Accelerated Dosing Regimen (LADR) Protocol: Pre-Transplant Treatment to Prevent Recurrence of Hepatitis C Virus (HCV) After Liver Transplantation
Brief Title: Pre-Transplant Treatment to Prevent Recurrence of Hepatitis C After Liver Transplantation
Acronym: LADR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: Schering-Plough (Industry); Ortho Biotech Clinical Affairs, L.L.C. (Industry)
Responsible Party: Principal Investigator, Averell Sherker, Division of Digestive Diseases and Nutrition, National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A2ALL LADR Protocol 62498(IND); U01DK062498 (NIH); U01DK062536 (NIH); U01DK062444 (NIH); U01DK062467 (NIH); U01DK062483 (NIH); U01DK062484 (NIH); U01DK062494 (NIH); U01DK062496 (NIH); U01DK062505 (NIH); U01DK062531 (NIH); CRADA through NIH-NIDDK (Other: Schering-Plough); CTA through NIH-NIDDK (Other: Ortho-Biotech); HRSA (Other: Health Resources and Services Administration); ASTS (Other: American Society of Transplant Surgeons)
Record Dates: First submitted 2005-08-24; First posted 2005-08-26 (Estimated); Results first posted 2013-04-04 (Estimated); Last update posted 2013-04-23 (Estimated); Status verified 2013-04

CONDITIONS: Hepatitis C
Keywords: Hepatitis C; Ribavirin; PegInterferon alfa2b
MeSH Terms: conditions — Hepatitis C | interventions — peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- LADR Treatment, Genotypes 1,4,6 (Experimental): Subjects randomized to low accelerating dose regimen (LADR) treatment
  Interventions: Drug: LADR Treatment
- Standard care (No Intervention): Subjects randomized to Standard Care group, Genotypes 1,4,6
- LADR treatment, Genotypes 2,3 (Experimental): Subjects randomized to low accelerating dose regimen (LADR) treatment.
  Interventions: Drug: LADR Treatment

INTERVENTIONS:
Drug: LADR Treatment — PEG-Intron (peginterferon alfa-2b (PEGIFN)) Redipen; Rebetol (ribavirin (RBV) United States Pharmacopeia (USP)) Capsules:
  Treatment was initiated with PEGIFN 0.75 µg/kg/week and RBV 600 mg/day. Dose escalations were performed at weeks 1 (PEGIFN 1.5 µg/kg/week and RBV 800 mg/day), 2 (RBV 1.0 g/day), and 3 (RBV 1.2 g/day for patients who weighed more then 75 kg) based upon patient tolerance and weekly blood counts. Once a patient reached the target RBV dose of 1-1.2 g/day (approximately 10.6 to 13.2 mg/kg/day), no further increases in RBV dose were made. Subsequent doses of PEGIFN and RBV were adjusted based upon adverse events, patient tolerability, and blood counts. If the highest tolerated dose of PEGIFN was <0.5 ug/kg, PEGIFN was permanently discontinued.
  Other Names: PEG-Intron; Rebetol; Low Accelerated Dosing Regimen
  Arms: LADR Treatment, Genotypes 1,4,6; LADR treatment, Genotypes 2,3

SUMMARY:
The purpose of this study is to learn if pre-liver transplant treatment, using peginterferon plus ribavirin, will clear hepatitis C virus (HCV) RNA from the blood in HCV-infected recipients and reduce the risk of recurrent HCV and allograft hepatitis following liver transplant.

DETAILED DESCRIPTION:
Patients awaiting deceased donor liver transplant will be asked to enroll in this protocol at the time of identification of a potential living liver donor (see note note at end of description). Patients randomized to treatment arm will be encouraged to delay living donor liver transplant (LDLT) until they have received 12 weeks of treatment to allow for a treatment response, if any, to occur. The pros and cons of immediate versus delayed LDLT will be discussed with each patient; the timing of LDLT for patients randomized to no treatment will be determined by clinical need. There will be separate treatment strategies depending upon HCV genotype. Preliminary data and experience strongly suggests that interferon-based treatment clears HCV RNA in the majority of patients with genotypes 2 and 3, even at lower than standard doses (79% on-treatment response and 50% SVR). In contrast, clearance rates for genotype 1 patients with advanced cirrhosis may only be 28% on-treatment with an 11% SVR. In addition, treatment may be associated with significant side effects, intolerance, and increased risk of complications of liver disease. The HCV Committee for A2ALL strongly agreed that monitoring safety of pre-transplant antiviral therapy was essential and advised inclusion of an untreated control group. For these reasons, all patients with HCV, genotypes 1, 4, 5, & 6 infection will be randomized 2:1 to either treatment or control (no treatment). Randomization will be web-based to avoid prior knowledge of treatment assignment at any site. In contrast to the randomized design for patients with genotypes 1, 4, 5, and 6, all patients with genotypes 2 and 3 HCV will receive treatment. All genotypes will be included in the analysis of safety, tolerance, and complications occurring during pre-transplant treatment.

Treatment is continued up to the time of LDLT or deceased donor liver transplant (DDLT), or to a maximum of 48 weeks of continuous treatment. Both peginterferon and ribavirin will be stopped if transplantation is expected to occur within 24 hours. Patients whose liver disease stabilize and are no longer in need of a liver transplant will complete a full 48 weeks of treatment with the aim of achieving SVR. These patients will be followed by measurement of HCV RNA, biochemical tests, hematology, and clinical evaluation at 3, 6, and 12 months post-treatment. If relapse occurs when treatment is discontinued after 48 weeks of therapy, institution of retreatment will be at the discretion of the investigator.

Deferral of LDLT while antiviral therapy is continued will be considered in patients who have undetectable HCV RNA, tolerate treatment well, lack evidence of HCC or ongoing hepatic decompensation, and have had stabilization or improvement in clinical or biochemical measures of liver disease: Child-Turcotte-Pugh (CTP) and Model for End-stage Liver Disease (MELD) scores. These patients should lack uncontrolled or ongoing bleeding from portal hypertension, ascites, systolic blood pressure (SBP), or encephalopathy. The decision to defer transplantation and to continue antiviral therapy will be made at the transplant center by the clinical investigator in consultation with the patient.

Based upon the kinetics of early virologic response in the peginterferon + ribavirin clinical trials, the researchers anticipate that a minimum of 12 weeks treatment is necessary to achieve a virologic response. However, the optimum duration of pre-transplant antiviral therapy that yields the highest rates of prevention of post-transplant HCV recurrence is unknown. Prolongation of antiviral therapy beyond 12 weeks may be advantageous in this regard, but prolonged therapy may also increase the risk of development of intercurrent complications of liver disease or side effects of treatment. In addition, patients with stable liver disease who achieve virologic remission may experience hepatic improvement and avoid transplantation.

All patients, treated and untreated controls will be followed and tested at the same intervals unless specified. Unscheduled visits and additional tests may be performed if clinically indicated, the findings at these visits and results of additional tests will be recorded in the database. The following details the schedule of visits and the tests/procedures to be performed at each visit:

Baseline

* History and Physical Examination
* Vital signs: Weight, blood pressure (BP), heart rate (HR), Temperature
* Fundoscopic exam in all patients. In patients with hypertension or diabetes exam should be performed with pupils dilated
* Quality of Life and Depression Assessment (SF-36V2, Beck Depression Inventory)
* Functional status evaluation
* Symptom assessment
* HCV RNA
* HCV Genotype
* Urinalysis
* Pregnancy Test
* HIV Test
* Other blood tests, including: complete blood count (CBC), International Normalized. Ratio (INR), Liver Panel, Creatine, Sodium Alpha-fetoprotein, triglycerides, iron studies, uric acid, thyroid stimulating hormone (TSH), antinuclear antibody (ANA)
* Ultrasound (US), computed tomography (CT), and/or magnetic resonance imaging (MRI) (some or all are probably done in LDLT evaluation)

Week 0 (Randomization and/or Treatment Start)

* Confirm eligibility
* Initiate treatment for all genotype 2, 3 patients and genotype 1, 4, 5 or 6 patients randomized to treatment group
* Repeat CBC, chemistries, INR

After randomization

* Week 1 and 3: CBC (for treated patients only, may be performed in local labs)
* Every 2 weeks up to 12 weeks: CBC, chemistries
* Weeks 4 and 8: Focused physical exam (signs and symptoms of liver disease) vital signs, urinalysis and symptom assessment
* Every 4 weeks from 12 to 48 weeks: Full physical exam and vital signs, urinalysis and symptom assessment, CBC, chemistries.
* Every 12 weeks up to 48 weeks: INR, TSH, urine or serum pregnancy test female (treated subjects of childbearing capacity only)
* At 12 Weeks: HCV RNA is measured. Patients without a 2-log or more drop in HCV RNA level are declared nonresponders and treatment is discontinued.
* After 12 weeks: HCV RNA is measured every 12 weeks on treatment by quantitative tests.
* At the time of LDLT or DDLT: CBC, INR, chemistries, quantitative and qualitative HCV RNA, Medications, adverse events (AE)
* Blood samples will be collected at Treatment Weeks 4, 8, 12, 24, 48 and at time of transplantation for subsequent HCV RNA testing in a central lab
* Quality of life (QOL) assessment at week 12, 24 and 48: Beck Depression Inventory (BDI) and SF-36V2
* Patients who discontinue treatment early due to adverse events will be followed according to the study schedule until 12 months after transplant or 48 weeks after randomization.

Post-LT (LDLT or DDLT) Follow-up

* Week 12, 24 and 52: CBC, INR, chemistries, HCV RNA by quantitative testing (part of A2ALL prospective study)
* Week 12, 24 and 52: Full physical exam and vital signs, urinalysis and symptom assessment
* Week 12: TSH and urine or serum pregnancy test (treated subjects of childbearing capacity only)
* Week 12, 24 and 52: QOL Assessment (BDI, and SF-36V2)
* Week 12 and 52: Liver Biopsy (part of A2ALL prospective study). Pathologists reading the 3 and 12 month biopsies will be blinded to the patients' clinical course and treatment.
* Blood samples will be collected at Week 12, 24 and 52 for subsequent HCV RNA testing in a central laboratory

Follow-up of Patients completing 48 weeks of Treatment without Transplantation

* Week 12, 24 and 48: CBC, INR, chemistries, HCV RNA by quantitative testing
* Week 12, 24 and 48: Full physical exam and vital signs, urinalysis and symptom assessment
* Week 12: TSH and urine or serum pregnancy test (treated subjects of childbearing capacity only)
* Week 12, 24 and 48: QOL Assessment (BDI, and SF-36V2)
* Blood samples will be collected at Week 12, 24 and 48 for subsequent HCV RNA testing in a central laboratory

NOTE: As a result of LADR Protocol Amendment III, patients with hepatocellular carcinoma (HCC) and tumor stage T2 awaiting DDLT are now eligible to participate in the LADR study. The following inclusion criteria was added:

• Candidates for DDLT who are listed for transplantation and meet United Network for Organ Sharing (UNOS) criteria for MELD upgrade for HCC

HCC DDLT candidates will not have their transplant delayed if a liver becomes available even if they have not completed 12 weeks of Rx.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18 or older)
* LDLT candidate
* HCV RNA positive
* Expected time on treatment is at least 12 weeks
* Candidates for DDLT who are listed for transplantation and meet UNOS criteria for MELD upgrade for HCC

Exclusion Criteria:

* Severe cytopenia (polymorphonuclear (PMN) leukocytes < 750, OR hemoglobin [Hgb] < 10 g/dL, OR platelet count < 35,000/mm3)
* Uncontrolled depression or psychiatric disease characterized by current symptoms of major depression or other psychiatric disease or increase in medication for major depression or other psychiatric disease within the past three months.
* Uncontrolled cardiopulmonary disease characterized by myocardial infarction, coronary artery bypass graft surgery, Percutaneous coronary intervention, or unstable angina within the past three months.
* Uncontrolled autoimmune disease characterized by current symptoms of autoimmune disease or increase in medications within the last three months.
* Autoimmune hepatitis
* Active substance abuse within 6 months of initiation of treatment
* Known intolerance or serious adverse event during prior therapy with interferon or ribavirin
* Prior nonresponse after at least 24 weeks of full dose treatment with peginterferon plus ribavirin
* Laboratory Model for End-Stage Liver Disease (MELD) score >20. Patients with laboratory MELD score 21-25 may be enrolled if deemed appropriate by the site investigator
* Serum creatinine >2.2 mg/dL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2005-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory T. Everson, MD, Study Chair — University of Colorado, Denver; James Everhart, MD, Study Director — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (8):
- United States (8):
  - University of California Los Angeles, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - University of Colorado, Denver, Colorado
  - Northwestern University Division of Transplantation, Chicago, Illinois
  - Columbia University, New York, New York
  - University of Pennsylvania Hospital, Philadelphia, Pennsylvania
  - University of Virginia, Charlottesville, Virginia
  - Virginia Commonwealth University, Richmond, Virginia

REFERENCES:
- [Background] Everson GT, Trotter J, Forman L, Kugelmas M, Halprin A, Fey B, Ray C. Treatment of advanced hepatitis C with a low accelerating dosage regimen of antiviral therapy. Hepatology. 2005 Aug;42(2):255-62. doi: 10.1002/hep.20793. PMID 16025497
- [Background] Stravitz RT, Shiffman ML, Sanyal AJ, Luketic VA, Sterling RK, Heuman DM, Ashworth A, Mills AS, Contos M, Cotterell AH, Maluf D, Posner MP, Fisher RA. Effects of interferon treatment on liver histology and allograft rejection in patients with recurrent hepatitis C following liver transplantation. Liver Transpl. 2004 Jul;10(7):850-8. doi: 10.1002/lt.20189. PMID 15237368
- [Background] Fried MW, Shiffman ML, Reddy KR, Smith C, Marinos G, Goncales FL Jr, Haussinger D, Diago M, Carosi G, Dhumeaux D, Craxi A, Lin A, Hoffman J, Yu J. Peginterferon alfa-2a plus ribavirin for chronic hepatitis C virus infection. N Engl J Med. 2002 Sep 26;347(13):975-82. doi: 10.1056/NEJMoa020047. PMID 12324553
- [Background] Manns MP, McHutchison JG, Gordon SC, Rustgi VK, Shiffman M, Reindollar R, Goodman ZD, Koury K, Ling M, Albrecht JK. Peginterferon alfa-2b plus ribavirin compared with interferon alfa-2b plus ribavirin for initial treatment of chronic hepatitis C: a randomised trial. Lancet. 2001 Sep 22;358(9286):958-65. doi: 10.1016/s0140-6736(01)06102-5. PMID 11583749
- [Result] Everson GT, Terrault NA, Lok AS, Rodrigo del R, Brown RS Jr, Saab S, Shiffman ML, Al-Osaimi AM, Kulik LM, Gillespie BW, Everhart JE; Adult-to-Adult Living Donor Liver Transplantation Cohort Study. A randomized controlled trial of pretransplant antiviral therapy to prevent recurrence of hepatitis C after liver transplantation. Hepatology. 2013 May;57(5):1752-62. doi: 10.1002/hep.25976. Epub 2013 Jan 17. PMID 22821361

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Persons were enrolled from October 2005 to January 2009, and followed through December 2009. Patients were enrolled at 7 clinical transplant centers in the United States.
Pre-assignment Details: No pre-assignment events. Randomization occurred immediately after enrollment.
Groups:
- Standard Clinical Care: Genotypes 1, 4, 6: Subjects randomized to non-treatment group 1:2 compared to treatment group.
- LADR Treatment: Genotypes 1, 4, 6: Low Accelerating Dose Regimen (LADR): Subjects randomized to LADR treatment group 2:1 compared to standard care.
- LADR Treatment: Genotypes 2 or 3: Patients in this subgroup were all assigned to LADR treatment.
Period: Overall Study
Arm/Group | Standard Clinical Care: Genotypes 1, 4, 6 | LADR Treatment: Genotypes 1, 4, 6 | LADR Treatment: Genotypes 2 or 3
Started | 16 | 31 | 32
Completed | 16 | 31 | 32
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Clinical Care: Genotypes 1, 4, 6 | LADR Treatment: Genotypes 1, 4, 6 | LADR Treatment: Genotypes 2 or 3 | Total
Number analyzed (Participants) | 16 | 31 | 32 | 79
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 15 | 30 | 27 | 72
  >=65 years | 1 | 1 | 5 | 7
Age Continuous [Mean (Standard Deviation); unit: years] | 56.1 (5.4) | 54.6 (7.4) | 56.6 (6.5) | 55.7 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 10 | 7 | 20
  Male | 13 | 21 | 25 | 59
Region of Enrollment [Number; unit: participants]
  United States | 16 | 31 | 32 | 79

OUTCOME MEASURES:

1. Primary Outcome: Patients Who Are Negative for Hepatitis C Virus (HCV) RNA at 3 Months Post-transplant: Intent-to-Treat Analysis (ITT)
Description: Post-transplant virologic response (pTVR) defined as undetectable HCV RNA at week 12 after liver transplantation.
Time Frame: 3 months post-transplant
Population: Intent-to-Treat (ITT) analyses of Transplanted patients assigned to treatment. Outcome is pTVR (post-transplant viral response)
Measure: Number; unit: participants
Groups:
- Standard Care Group: Genotypes 1, 4, 6; LADR Treatment Group: Genotypes 1, 4, 6: Randomization 2:1 LADR vs. Standard care in Genotypes 1,4,6
- LADR Treatment Group: Genotypes 2, 3: All patients with Genotypes 2,3 received LADR treatment.
Arm/Group | Standard Care Group: Genotypes 1, 4, 6 | LADR Treatment Group: Genotypes 1, 4, 6 | LADR Treatment Group: Genotypes 2, 3
Number analyzed (Participants) | 13 | 24 | 22
participants | 0 [lower limit 0] | 5 [0.07 to 0.42] | 6 [0.11 to 0.50]
Statistical Analysis 1: Comparison: Standard Care Group: Genotypes 1, 4, 6 vs LADR Treatment Group: Genotypes 1, 4, 6 vs LADR Treatment Group: Genotypes 2, 3; ITT analysis of pTVR: 0/13 Standard care vs. 11/46 Combined LADR-treated groups; Test type: Superiority or Other; p = 0.0477, Fisher Exact — One-sided test
Statistical Analysis 2: Comparison: LADR Treatment Group: Genotypes 1, 4, 6 vs LADR Treatment Group: Genotypes 2, 3; ITT analysis of LADR-treated: 5/24 Genotypes 1,4,6 vs 6/22 Genotypes 2,3; Test type: Superiority or Other; p = 0.6090, Chi-squared

2. Secondary Outcome: Patients With Combined Virologic Response (CVR): Intent-to-Treat Analyses (ITT)
Description: Intent-to-Treat (ITT) analyses of all patients. Combined Virologic Response (CVR), which includes both sustained virologic response pre-transplant (SVR) and post-transplant virologic response (pTVR)
Time Frame: Pre-transplant and 3 months post-transplant
Population: All study patients
Measure: Number; unit: participants
Arm/Group | Standard Care Group: Genotypes 1, 4, 6 | LADR Treatment Group: Genotypes 1, 4, 6 | LADR Treatment Group: Genotypes 2, 3
Number analyzed (Participants) | 16 | 31 | 32
participants | 1 | 6 | 6
Statistical Analysis 1: Comparison: Standard Care Group: Genotypes 1, 4, 6 vs LADR Treatment Group: Genotypes 1, 4, 6 vs LADR Treatment Group: Genotypes 2, 3; ITT analysis of CVR: 1/16 Standard care vs. 12/63 Combined LADR-treated groups; Test type: Superiority or Other; p = 0.2014, Fisher Exact — One-sided test
Statistical Analysis 2: Comparison: LADR Treatment Group: Genotypes 1, 4, 6 vs LADR Treatment Group: Genotypes 2, 3; ITT analysis of LADR-treated: 6/31 Genotypes 1,4,6 vs 6/32 Genotypes 2,3; Test type: Superiority or Other; p = 0.9513, Chi-squared

3. Primary Outcome: Patients Who Are Negative for HCV RNA at 3 Months Post-transplant: Per-Protocol Analysis (PP)
Description: Post-transplant virologic response (pTVR) defined as undetectable HCV RNA at week 12 after liver transplantation, analysed among patients who received treatment.
Time Frame: 3 months post-transplant
Population: Per-Protocol (PP) analyses of Transplanted patients who received treatment. Outcome is pTVR (post-transplant viral response)
Measure: Number; unit: participants
Arm/Group | Standard Care Group: Genotypes 1, 4, 6 | LADR Treatment Group: Genotypes 1, 4, 6 | LADR Treatment Group: Genotypes 2, 3
Number analyzed (Participants) | 13 | 23 | 21
participants | 0 | 5 | 6
Statistical Analysis 1: Comparison: Standard Care Group: Genotypes 1, 4, 6 vs LADR Treatment Group: Genotypes 1, 4, 6 vs LADR Treatment Group: Genotypes 2, 3; PP analysis of pTVR: 0/13 Standard care vs. 11/44 Combined LADR-treated groups; Test type: Superiority or Other; p = 0.0274, Fisher Exact — One-sided test
Statistical Analysis 2: Comparison: LADR Treatment Group: Genotypes 1, 4, 6 vs LADR Treatment Group: Genotypes 2, 3; PP analysis of LADR-treated: 5/23 G1,4,6 vs 6/21 G2,3; Test type: Superiority or Other; p = 0.6011, Chi-squared

4. Secondary Outcome: Patients With Combined Virologic Response (CVR): Per-Protocol Analysis (PP)
Description: Per-Protocol (PP) analyses of all patients. Combined Virologic Response (CVR)includes both sustained virologic response pre-transplant (SVR) and post-transplant virologic response (pTVR), analysed among patients who received treatment.
Time Frame: Pre-transplant and 3 months post-transplant
Population: All study patients
Measure: Number; unit: participants
Arm/Group | Standard Care Group: Genotypes 1, 4, 6 | LADR Treatment Group: Genotypes 1, 4, 6 | LADR Treatment Group: Genotypes 2, 3
Number analyzed (Participants) | 20 | 30 | 29
participants | 0 | 7 | 6
Statistical Analysis 1: Comparison: Standard Care Group: Genotypes 1, 4, 6 vs LADR Treatment Group: Genotypes 1, 4, 6 vs LADR Treatment Group: Genotypes 2, 3; PP analysis of CVR: 0/20 Standard care vs. 13/59 Combined LADR-treated groups; Test type: Superiority or Other; p = 0.0153, Fisher Exact — One-sided test
Statistical Analysis 2: Comparison: LADR Treatment Group: Genotypes 1, 4, 6 vs LADR Treatment Group: Genotypes 2, 3; PP analysis of LADR-treated: 7/30 G1,4,6 vs 6/29 G2,3; Test type: Superiority or Other; p = 0.8065, Chi-squared

ADVERSE EVENTS:
Time Frame: Serious Adverse Events (SAE) were collected pre-transplant, and through 1 year post-transplant.
Description: Other [non-serious] adverse events were not collected or assessed as part of this study.
Groups:
- Standard Clinical Care: Genotypes 1, 4, 6: Subjects who received no LADR treatment (Per Protocol analysis)
- LADR Treatment (All Genotypes): This group combines all who received LADR treatment (Per Protocol analysis) for all Genotypes 1,4,6 and 2,3
Arm/Group | Standard Clinical Care: Genotypes 1, 4, 6 | LADR Treatment (All Genotypes)
Serious Adverse Events (participants affected / at risk) | 11/20 | 40/59
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Standard Clinical Care: Genotypes 1, 4, 6 (N=20) | LADR Treatment (All Genotypes) (N=59)
Death (General disorders) | 2 (2) | 9 (9)
Pre-LT Cytopenia (Blood and lymphatic system disorders) | 0 (0) | 8 (11)
Pre-LT Infection (Infections and infestations) | 0 (0) | 3 (7)
Pre-LT Liver-related (Hepatobiliary disorders) | 3 (3) | 6 (8)
Pre-LT Other (General disorders) | 1 (1) | 10 (11)
Post-LT (first 30 days) Cytopenia (Blood and lymphatic system disorders) | 0/13 (0) | 0/44 (0)
Post-LT (first 30 days) Infection (Infections and infestations) | 0/13 (0) | 3/44 (4)
Post-LT (first 30 days) Liver-related (Hepatobiliary disorders) | 1/13 (1) | 3/44 (3)
Post-LT (first 30 days) Rejection (Hepatobiliary disorders) | 0/13 (0) | 1/44 (1)
Post-LT (first 30 days) Surgical complication (Surgical and medical procedures) | 0/13 (0) | 1/44 (2)
Post-LT (first 30 days) Other (General disorders) | 1/13 (1) | 6/44 (7)
Post-LT (30 days-1 year) Cytopenia (Blood and lymphatic system disorders) | 1/13 (2) | 0/44 (0)
Post-LT (30 days-1 year) Infection (Infections and infestations) | 3/13 (3) | 7/44 (9)
Post-LT (30 days-1 year) Liver-related (Hepatobiliary disorders) | 0/13 (0) | 1/44 (2)
Post-LT (30 days-1 year) Rejection (Hepatobiliary disorders) | 0/13 (0) | 0/44 (0)
Post-LT (30 days-1 year) Surgical complication (Surgical and medical procedures) | 0/13 (0) | 6/44 (8)
Post-LT (30 days-1 year) Other (General disorders) | 2/13 (2) | 10/44 (13)

LIMITATIONS AND CAVEATS:
Failure to reach target of 84 transplanted patients (47 achieved); Inability to complete planned 12 weeks of treatment for some; Incomplete HCV RNA follow up; Inconsistent limits of detection of HCV RNA; Noncompliance with assigned treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No